CLINICAL TRIAL: NCT06414564
Title: Effects of Advanced Hybrid Closed-loop System on Glycemic Control and Psychosocial Outcomes in Pediatric Patients With Type 1 Diabetes
Brief Title: Effects of AHCL Insulin Pump on Glycemic Control and Psychosocial Outcomes in Pediatric Patients With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Lee Young Ah, Associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23081591461
Record Dates: First submitted 2024-01-30; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AHCL system application (Experimental): insulin infusion using AHCL system insulin pump (Medtronic 780G) with continous glucose monitoring (guardian G4)
  Interventions: Device: Medtronic 780G insulin pump

INTERVENTIONS:
Device: Medtronic 780G insulin pump — Subjects on insulin infusion by 780G AHCL system

SUMMARY:
Prospective, non-randomized, single-arm clinical trial to investigate the effects of advanced hybrid close-loop (AHCL) system insulin pump in pediatric patients with type 1 diabetes

DETAILED DESCRIPTION:
This trial consists of baseline phase of 3 weeks sustaining the treatment previously maintained by the patient, followed by study phase of 12 weeks of AHCL system application.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is age 7-19
2. The subject with one or more of the below

   * serum c-peptide ≤ 0.6 ng/mL at diagnosis
   * positive glutamic acid decarboxylase (GAD) antibody
   * positive islet cell antibody
   * positive anti-Insulin antibody
   * positive anti-islet Antigen-2 (IA-2) antibody
3. The subject was diagnosed with type 1 diabetes ≥ 1 year
4. The subject has been continuously treated at least for 8 weeks at the start of the study, by one of the existing insulin treatment methods [insulin multi-injection (MDII), general insulin pump (CSII), sensor-linked insulin pump (SAP), or 770G insulin pump (HCL system)]
5. The subject has been applied with real-time continuous glucose monitoring at least for 8 weeks at the start of the study

Exclusion Criteria:

1. Any systemic treatment with drugs known to interfere with glucose metabolism within 8 weeks prior to trial
2. Subjects with underlying hematologic disorders that can affect the HbA1c levels
3. Subjects with underlying medical disorders that can affect glucose metabolism
4. Subjects with a neuropsychiatric disorder such as depression or eating disorder
5. Subjects with underlying thyroid disorders and abnormal thyroid function

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time In Range (TIR) | baseline (3 weeks) and intervention (12 weeks) period
  glucose level between 70-180 mg/dL derived from continuous glucose monitoring

SECONDARY OUTCOMES:
Time Above Range (TAR) | baseline (3 weeks) and intervention (12 weeks) period
  glucose level >180 mg/dL derived from continuous glucose monitoring
Time Below Range (TBR) | baseline (3 weeks) and intervention (12 weeks) period
  glucose level <70 mg/dL derived from continuous glucose monitoring
mean sensor glucose | baseline (3 weeks) and intervention (12 weeks) period
  mean sensor glucose level derived from continuous glucose monitoring
Coefficient of variation (CV) | baseline (3 weeks) and intervention (12 weeks) period
  Standard deviation * 100/ mean (derived from continuous glucose monitoring)
Glucose management indicator (GMI) | baseline (3 weeks) and intervention (12 weeks) period
  Estimated HbA1c levels derived from continuous glucose monitoring
HbA1c | before and at the end of intervention, which in average lasts 12 weeks
  Glycated hemoglobin level
Glycated albumin | before and at the end of intervention, which in average lasts 12 weeks
  Glycated albumin level
Quality of life measurements (general) of patients and parents | baseline (3 weeks) and intervention (12 weeks) period
  Measured by PedsQL (Pediatric Quality of Life InventoryTM) Generic Core, Module 4.0 (values: 0~100, higher score means better outcome)
Quality of life measurements (diabetes-specific) of patients and parents | baseline (3 weeks) and intervention (12 weeks) period
  Measured by PedsQL (Pediatric Quality of Life InventoryTM) Diabetes Specific, Module 3.0 (values: 0~100, higher score means better outcome)
Children's Depression Inventory(CDI) (age 7-17) or Beck Depression Inventory (BDI) (age 18-19) of patients | baseline (3 weeks) and intervention (12 weeks) period
  Measured by Korean Children's Depression Inventory, 2nd Edition (values: 0~100, higher score means worse outcome) or Korean Beck Depression Inventory, 2nd Edition (higher score means worse outcome)

OTHER OUTCOMES:
Sleep enter and end time | baseline (3 weeks) and intervention (12 weeks) period
  Measured in time, derived from Fitbit data
Sleep duration | baseline (3 weeks) and intervention (12 weeks) period
  Measured in hours and minutes, derived from Fitbit data
Sleep efficiency | baseline (3 weeks) and intervention (12 weeks) period
  Derived from Fitbit data
Wake after sleep onset | baseline (3 weeks) and intervention (12 weeks) period
  Derived from Fitbit data

CONTACTS AND LOCATIONS:
Overall Officials: Young Ah Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea